CLINICAL TRIAL: NCT01278498
Title: A Multicenter, Double Blind Trial to Compare the Efficacy and Safety of Escitalopram With Placebo in Patients With Acute Stroke for the Prevention of Poststroke Depression and Related Symptoms (Emotional Incontinence, Anger Proneness), and for Improvement of Neurologic, Cognitive Function and Quality of Life
Brief Title: The Preventive Effect of Escitalopram on Depression and Related Emotional Disorders in Acute Stroke Patients
Acronym: EMOTION
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Dong-A ST Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jongsung Kim, professor, department of neurology, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EMOTION
Record Dates: First submitted 2011-01-18; First posted 2011-01-19 (Estimated); Last update posted 2014-10-09 (Estimated); Status verified 2014-10

CONDITIONS: Depression
Keywords: Escitalopram; Depression; Stroke
MeSH Terms: conditions — Depression; Stroke | interventions — Escitalopram; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- escitalopram (Experimental): prevention of poststroke depression in patients with acute stroke.
  Interventions: Drug: Escitalopram
- placebo (Placebo Comparator): prevention of poststroke depression in patients with acute stroke.
  Interventions: Drug: sugar pill

INTERVENTIONS:
Drug: Escitalopram — first week:5mg 2nd week~12 week:10mg
  Other Names: lexacure
  Arms: escitalopram
Drug: sugar pill — first week:5mg 2nd week~12 weeks:10mg
  Other Names: Placebo
  Arms: placebo

SUMMARY:
Through this study, the investigators are to demonstrate the superiority of Escitalopram over placebo for the prevention of poststroke depression in patients with acute stroke

The primary hypothesis of this study is;

This study will prove the superiority of Escitalopram on the prevention of poststroke depression in patients with acute stroke against placebo

DETAILED DESCRIPTION:
This study is to randomize stroke patients either to the SSRI, Lexacure tablet or placebo and to investigate whether Lexacure is effective in preventing depression and related symptoms at 3 months after the drug administration.

Patients with acute stroke (within 21 days after onset) will be enrolled and take the study drug 5mg during the first week and then 10mg (from the 2nd week) until 12 weeks.

The first visit should be performed at 4 weeks after drug administration. Drug safety, depression and related symptoms will be evaluated and the following 12-week visit will be performed. In the 13th week after the drug administration, the study drug will be reduced to 10mg every other day for one week, and the schedule of drug administration will be completed.

At the 14th week, all subjects will be instructed not to take the study drug for assessing maintenance effect. At the 24th week, subjects will have follow-up visits to assess poststroke depression and related symptoms.

If a subject discontinues the study before termination for severe depression, aggressive intervention will be initiated at the 4th week, and the 12-week visit will be performed unless the subject disagrees. If investigators judge the patients have severe depression at the 12-week visit, they should be treated. All the patients who need to treat depression will be followed until 12th week.

ELIGIBILITY:
Inclusion Criteria:

* Adults older than 20 years
* Patients with acute stroke (ischemic stroke or cerebral hemorrhage) confirmed by neuroimaging within 21 days after stroke onset
* Patients with hemorrhagic transformation of infarcted tissue will not be included, but if investigators judge the risk of bleeding is small (i.e., reduced amount of blood in follow-up neuroimaging) those patients can be enrolled.
* Patients with MRS ≥ 2 on screening
* Patients without definite history of depression
* Patients who fulfill the following criteria in the K-MADRS test:

The combined score of the 9th question (pessimistic thoughts) and the 10th question (suicidal idea) ≤ 7 The score of the 10th question < 6

* Patients without serious communication problem
* Patients who agree to participate in this trial

Exclusion Criteria:

* Patients with MRS 0 or 1 on screening
* Patients who have definite history of depression or have taken antidepressants
* Patients who have been diagnosed as having bipolar disorder or other psychiatric disorders
* Patients with severe dementia or aphasia. However, those who have motor aphasia but are still communicable can be enrolled
* Patients who have taken migraine medication on screening or those who are expected to take migraine medication frequently due to severe migraine
* Patients who have strong suicidal idea on screening test or those who express their wish to be treated for depression
* Patients who are considered to be treated for depression by charged physicians
* Patients who need SSRI medication for other reasons
* Patients who have taken antiepileptic drugs on screening
* Patients who have a history of traumatic brain injury, brain tumor, or other brain disease (except stroke) within 30 days prior to screening
* Patients with uncommon causes of stroke (e.g. subarachnoid hemorrhage, venous thrombosis, arteriovenous malformation, or Moyamoya disease)
* Patients with bleeding diathesis, hemophilia, or thrombocytopenia
* Patients with severe concomitant illness (e.g. liver disease, renal disease, malignancy)
* Patients with abnormal blood tests Abnormal LFT (ALT > 200 or AST > 200) Anemia (Hb < 8 mg/dl) or thrombocytopenia (<100,000/mm3) Renal insufficiency (Cr > 3.0 mg/dl) or renal failure requiring dialysis Patients with severe heart failure (NYHA class III or IV) NYHA classification for heart failure Class I : patients with no limitation of activities; they suffer no symptoms from Ordinary activities Class II : patients with slight, mild limitation of activity; they are comfortable with rest or with mild exertion Class III : patients with marked limitation of activity; they are comfortable only at rest Class IV : patients who should be at complete rest, confined to bed or chair; any activity brings on
* Pregnant or lactating patients
* Patients who are participating in another clinical trial, but those who are participating in the observational study can be enrolled

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 444 (Estimated)
Dates: Start 2011-01; Primary Completion 2014-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Occurrence rate of depression | 3 months
  Occurrence rate of depression (Montgomery-Asberg Depression Scale score ≥16)

SECONDARY OUTCOMES:
Prevention of depression | 3 months
Prevention of emotional incontinence | 3, 6 months
Prevention of anger proneness | 3, 6 months
Recovery of neurologic dysfunction | 3, 6 months
Improvement of cognitive function | 3, 6 months
Improvement of quality of life | 3, 6 months
Improvement of caregiver burden | 3, 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jong Sung Kim, MD, PhD, Principal Investigator — Department of Neurology, Asan Medical Center
Locations (16):
- South Korea (16):
  - Kangwon National University Hospital, Chuncheon, Gangwon-do
  - Kwandong University College of Medicine Myongji Hospital, Gyeonggi-do, Goyang
  - Korea University Ansan Hospital, Ansan, Gyeonggi-do
  - Hanyang University Guri Hospital, Guri-si, Gyeonggi-do
  - Daegu Fatima Hospital, Daegu, Gyeongsang
  - Dongguk University International Hospital, Goyang, Kyoungki-do
  - Hallym Univesity Sacred Heart Hospital, Anyang
  - Dong-A University Hospital, Busan
  - Dongsan Medical Center, Daegu
  - Chungnam National University Hospital, Daejeon
  - Chosun University Hospital, Gwangju
  - Inha University Hospital, Inchon
  - Severance Hospital, Seoul
  - KyungHee University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Konkuk Univ. Hospital, Seoul

REFERENCES:
- [Derived] Lee EJ, Kim JS, Chang DI, Park JH, Ahn SH, Cha JK, Heo JH, Sohn SI, Lee BC, Kim DE, Kim HY, Kim S, Kwon DY, Kim J, Seo WK, Lee J, Park SW, Koh SH, Kim JY, Choi-Kwon S, Kim MS, Lee JS. Post-Stroke Depressive Symptoms: Varying Responses to Escitalopram by Individual Symptoms and Lesion Location. J Geriatr Psychiatry Neurol. 2021 Nov;34(6):565-573. doi: 10.1177/0891988720957108. Epub 2020 Sep 10. PMID 32912058
- [Derived] Lee EJ, Kim JS, Chang DI, Park JH, Ahn SH, Cha JK, Heo JH, Sohn SI, Lee BC, Kim DE, Kim HY, Kim S, Kwon DY, Kim J, Seo WK, Lee J, Park SW, Koh SH, Kim JY, Choi-Kwon S. Depressive Symptoms in Stroke Patients: Are There Sex Differences? Cerebrovasc Dis. 2020;49(1):19-25. doi: 10.1159/000506116. Epub 2020 Feb 5. PMID 32023608
- [Derived] Lee EJ, Kim JS, Chang DI, Park JH, Ahn SH, Cha JK, Heo JH, Sohn SI, Lee BC, Kim DE, Kim HY, Kim S, Kwon DY, Kim J, Seo WK, Lee J, Park SW, Koh SH, Kim JY, Choi-Kwon S, Kim MS, Lee JS; EMOTION Investigators. Differences in Therapeutic Responses and Factors Affecting Post-Stroke Depression at a Later Stage According to Baseline Depression. J Stroke. 2018 May;20(2):258-267. doi: 10.5853/jos.2017.02712. Epub 2018 May 31. PMID 29886724
- [Derived] Lee EJ, Oh MS, Kim JS, Chang DI, Park JH, Cha JK, Heo JH, Sohn SI, Kim DE, Kim HY, Kim J, Seo WK, Lee J, Park SW, Kim YJ, Lee BC; EMOTION investigators. Serotonin transporter gene polymorphisms may be associated with poststroke neurological recovery after escitalopram use. J Neurol Neurosurg Psychiatry. 2018 Mar;89(3):271-276. doi: 10.1136/jnnp-2017-316882. Epub 2017 Oct 13. PMID 29030421
- [Derived] Kim JS, Lee EJ, Chang DI, Park JH, Ahn SH, Cha JK, Heo JH, Sohn SI, Lee BC, Kim DE, Kim HY, Kim S, Kwon DY, Kim J, Seo WK, Lee J, Park SW, Koh SH, Kim JY, Choi-Kwon S; EMOTION investigators. Efficacy of early administration of escitalopram on depressive and emotional symptoms and neurological dysfunction after stroke: a multicentre, double-blind, randomised, placebo-controlled study. Lancet Psychiatry. 2017 Jan;4(1):33-41. doi: 10.1016/S2215-0366(16)30417-5. PMID 28012485